CLINICAL TRIAL: NCT01997411
Title: Assessment of Intranasal Glucagon in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Jaeb Center for Health Research (Other); Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16418; I8R-MC-IGBB (Other: Eli Lilly and Company); INGluc002 (Other: Jaeb Center for Health Research); AMG103 (Other: Locemia)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: IM and NG arms are open labeled. NG cohorts, 2mg and 3mg, are quadruple blinded.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Glucagon (NG) (Experimental): Nasal glucagon (NG) doses of 2.0 mg and 3.0 mg for participants 4 to less than 12 years of age and 3.0 mg for those 12 to less than 17 years of age were administered in a nostril with a prefilled delivery device that delivered a single dose upon activation.
  Interventions: Drug: Nasal Glucagon
- Intramuscular (IM) Glucagon (Active Comparator): Participants who weighed at least 25 kilograms (kg)/55 pounds (lbs) were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 lbs, IM glucagon dosed with 0.5 mg
  Interventions: Drug: Intramuscular Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon
  Other Names: AMG504-1; LY900018
  Arms: Nasal Glucagon (NG)
Drug: Intramuscular Glucagon
  Other Names: GlucaGen HypoKit
  Arms: Intramuscular (IM) Glucagon

SUMMARY:
The purpose of this study was to assess how glucagon administered nasally, using a nasal dosing delivery device, works in children and adolescents compared with commercially-available glucagon given by injection. In addition, the safety and tolerability of glucagon given nasally was evaluated.

DETAILED DESCRIPTION:
This study was conducted to permit determination of appropriate dose level(s) for pediatric use based on the safety observations and results of glucagon and glucose assays.

Each participant 12 to less than 17 years of age underwent two visits in random order and received glucagon nasal powder once and commercially available glucagon (GlucaGen, Novo Nordisk) by intramuscular (IM) injection once. Participants 4 to less than 12 years were randomly assigned to have either 1 visit with commercially available glucagon (GlucaGen, Novo Nordisk) by IM injection OR to have 2 visits with a 2.0 milligram (mg) dose of glucagon nasal powder administered during one visit and a 3.0 mg dose of glucagon nasal powder administered during the other visit. For those randomized to complete two research dosing visits, the dose of glucagon nasal powder given during each visit was masked to the participant and study personnel.

Glucagon was administered after glucose was lowered to <80 mg/dL using insulin if necessary on the dosing day. Participants were treated with either glucagon given nasally (either 2.0 mg or 3.0 mg for participants 4 to less than 12 years of age or 3.0 mg for those 12 to less than 17 years of age) or by intramuscular (IM) injection (1 mg for those 55 pounds [lbs] or more and 0.5 mg for those weighing less than 55 lbs) in the quadriceps muscle of the leg.

Blood glucose levels and adverse events were carefully monitored for 90 minutes post-dosing. After a wash-out period of 7 days or more, participants 12 to less than 17 years of age returned to the clinic and the procedure was repeated with each participant crossed over to the other treatment. Participants 4 to less than 12 years assigned to have 2 dosing visits returned to clinic for repeated procedures and received alternate dose of nasal glucagon (NG). Participants 4 to less than 12 years assigned to a single dosing visit did not return for a second dosing visit.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the following inclusion criteria were met:

* History of type 1 diabetes and receiving daily insulin therapy from the time of diagnosis for at least 12 months
* At least 4 years of age and less than 17 years
* Females must have met one of the following criteria:

  * Of childbearing potential but agreed to use an accepted contraceptive regimen as described in the study procedure manual throughout the entire duration of the study (from screening until study completion)
  * Of non-childbearing potential, defined as a female who had a hysterectomy or tubal ligation, was clinically considered infertile or had not yet reached menarche
* In good general health with no conditions that could have influenced the outcome of the trial, and in the judgment of the Investigator was a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
* Willingness to adhere to the study requirements

Exclusion Criteria:

An individual was not eligible if any of the following exclusion criteria were present:

* Females who were pregnant according to a positive urine pregnancy test, actively attempting to get pregnant, or were lactating
* History of hypersensitivity to glucagon or any related products or severe hypersensitivity reactions (such as angioedema) to any drugs
* Presence of cardiovascular, gastrointestinal, liver or kidney disease, or any other conditions which in the judgment of the investigator could have interfered with the absorption, distribution, metabolism or excretion of drugs or could potentiate or predispose to undesired effects
* History of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma
* History of an episode of severe hypoglycemia (as defined by an episode that required third party assistance for treatment) in the 1 month prior to enrolling in the study
* Use of daily systemic beta-blocker, indomethacin, warfarin or anticholinergic drugs
* History of epilepsy or seizure disorder
* Use of an Investigational Product in another clinical trial within the past 30 days
* Blood donation in 3 months prior to first glucagon dosing

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Riley Hospital for Children Indiana University Health, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - UPA Buffalo, Buffalo, New York

REFERENCES:
- [Derived] Sherr JL, Ruedy KJ, Foster NC, Piche CA, Dulude H, Rickels MR, Tamborlane WV, Bethin KE, DiMeglio LA, Fox LA, Wadwa RP, Schatz DA, Nathan BM, Marcovina SM, Rampakakis E, Meng L, Beck RW; T1D Exchange Intranasal Glucagon Investigators. Glucagon Nasal Powder: A Promising Alternative to Intramuscular Glucagon in Youth With Type 1 Diabetes. Diabetes Care. 2016 Apr;39(4):555-62. doi: 10.2337/dc15-1606. Epub 2016 Feb 16. PMID 26884472

RESULTS

PARTICIPANT FLOW:
Groups:
- 4 to<8 Years Old Intramuscular (IM) Glucagon Visit: Participants who weighed at least 25 kilograms (kg)/55 pounds (lbs) were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 Ibs, IM glucagon dose was 0.5 mg.
  This was completed at one visit and was the only visit for this cohort.
- 4 to <8 Years Old NG 2.0 mg 1st Visit/3.0 mg 2nd Visit: At the first visit, a nasal glucagon (NG) dose of 2.0 milligrams (mg) for participants 4 to less than 8 years of age was administered nasally.
  At the second visit, NG dose of 3.0 mg was administered nasally.
- 4 to <8 Years Old NG 3.0 mg 1st Visit/2.0 mg 2nd Visit: At the first visit, a NG dose of 3.0 mg for participants 4 to less than 8 years of age was administered nasally.
  At the second visit, a NG dose of 2.0 mg was administered nasally.
- 8 to <12 Years Old Intramuscular Glucagon Visit: Participants who weighed at least 25 kilograms kg/55 lbs were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 Ibs, IM glucagon dose was 0.5 mg. This was completed at one visit and was the only visit for this cohort.
- 8 to <12 Years Old NG 2.0 mg 1st Visit/3.0 mg 2nd Visit: At the first visit, a NG dose of 2.0 mg for participants 8 to less than 12 years of age was administered nasally.
  At the second visit, a NG dose of 3.0 mg was administered nasally.
- 8 to <12 Years Old NG 3.0 mg 1st Visit/2.0 mg 2nd Visit: At the first visit, a NG dose of 3.0 mg for participants 8 to less than 12 years of age was administered nasally.
  At the second visit, a NG dose of 2.0 mg was administered nasally.
- 12 to <17 Years Old NG 1st Visit/IM Glucagon 2nd Visit: At the first visit, a NG dose of 3.0 mg was administered nasally.
  At the second visit, participants who weighed at least 25 kg/55 lbs were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 Ibs, IM glucagon dose was 0.5 mg.
- 12 to <17 Years Old IM Glucagon 1st Visit/NG 2nd Visit: At the first visit, participants who weighed at least 25 kg/55 lbs were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 Ibs, IM glucagon dose was 0.5 mg.
  At the second visit, a NG dose of 3.0 mg was administered nasally.
Period: Overall Study
Arm/Group | 4 to<8 Years Old Intramuscular (IM) Glucagon Visit | 4 to <8 Years Old NG 2.0 mg 1st Visit/3.0 mg 2nd Visit | 4 to <8 Years Old NG 3.0 mg 1st Visit/2.0 mg 2nd Visit | 8 to <12 Years Old Intramuscular Glucagon Visit | 8 to <12 Years Old NG 2.0 mg 1st Visit/3.0 mg 2nd Visit | 8 to <12 Years Old NG 3.0 mg 1st Visit/2.0 mg 2nd Visit | 12 to <17 Years Old NG 1st Visit/IM Glucagon 2nd Visit | 12 to <17 Years Old IM Glucagon 1st Visit/NG 2nd Visit
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 4 to <8 Years Old IM Glucagon Cohort: Participants who were 4 to < 8 years old at the time of enrollment into the study randomized to receive only the intramuscular glucagon at one visit.
- 4 to <8 Years Old NG Cohort: Participants who were 4 to < 8 years old at the time of enrollment into the study randomized to receive 2.0 or 3.0 mg of nasal glucagon at two separate visits. Order of these visits was randomized.
- 8 to <12 Years Old IM Glucagon Cohort: Participants who were 8 to < 12 years old at the time of enrollment into the study randomized to receive only the intramuscular glucagon at one visit.
- 8 to <12 Years Old NG Cohort: Participants who were 8 to < 12 years old at the time of enrollment into the study randomized to receive 2.0 or 3.0 mg of nasal glucagon at two separate visits. Order of these visits was randomized.
- 12 to <17 Years Old NG/IM Cohort: Participants who were 12 to < 17 years old at the time of enrollment into the study randomized to receive either intramuscular glucagon or nasal glucagon at two separate visits. Order of these visits was randomized.
- Total: Total of all reporting groups
Arm/Group | 4 to <8 Years Old IM Glucagon Cohort | 4 to <8 Years Old NG Cohort | 8 to <12 Years Old IM Glucagon Cohort | 8 to <12 Years Old NG Cohort | 12 to <17 Years Old NG/IM Cohort | Total
Number analyzed (Participants) | 6 | 12 | 6 | 12 | 12 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.8 [5.7 to 7.5] | 6.8 [5.7 to 7.5] | 11.1 [10.5 to 11.8] | 11.1 [10.5 to 11.8] | 14.5 [13.2 to 15.8] | 10.6 [7.4 to 12.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 5 | 5 | 16
  Male | 6 | 9 | 3 | 7 | 7 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 12 | 6 | 12 | 12 | 48
Local HbA1c [Mean (Standard Deviation); unit: percent] | 7.6 (0.5) | 8.3 (0.8) | 7.5 (1.1) | 8.1 (0.7) | 8.2 (1.5) | 8.0 (1.0)
Duration of Diabetes [Median (Inter-Quartile Range); unit: years] | 3.1 [2.1 to 3.8] | 2.7 [1.8 to 3.6] | 5.3 [3.9 to 6.3] | 4.3 [3.4 to 6.7] | 5.9 [3.5 to 8.0] | 3.9 [2.6 to 6.0]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: All enrolled participants that completed the required dosing visit(s). One participant in the 4 to <8 year old 2.0 mg NG group was excluded due to blowing nose after NG administration. One participant in the 8 to <12 group withdrew after completion of the 3.0 mg NG visit and did not complete the 2.0 mg NG visit.
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Groups:
- 4 to<8 Years Old IM Glucagon Visit; 8 to <12 Years Old IM Glucagon Visit; 12 to <17 Years Old IM Glucagon Visit: Participants who weighed at least 25 kg/55 lbs were dosed 1 mg of IM glucagon; participants who weighed less than 25 kg/55 Ibs, IM glucagon dose was 0.5 mg.
- 4 to<8 Years Old NG Visit 2.0 mg: NG dose of 2.0 mg for participants 4 to less than 8 years of age.
- 4 to<8 Years Old NG Visit 3.0 mg: NG dose of 3.0 mg for participants 4 to less than 8 years of age.
- 8 to<12 Years Old NG Visit 2.0 mg: NG dose of 2.0 mg for participants 8 to less than 12 years of age.
- 8 to<12 Years Old NG Visit 3.0 mg: NG dose of 3.0 mg for participants 8 to less than 12 years of age.
- 12 to<17 Years Old NG Visit 3.0 mg: NG dose of 3.0 mg for participants 12 to less than 17 years of age.
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
picograms per millilitre (pg/mL) | 6290.33 (2045.96) | 3463.55 (1760.28) | 3958.58 (2438.60) | 4743.00 (3094.61) | 2776.27 (979.28) | 5664.33 (2114.69) | 4277.25 (3774.77) | 3103.25 (2302.61)

2. Primary Outcome: Time to Maximum Concentration (Tmax) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
hours (hr) | 0.29 [0.08 to 0.50] | 0.25 [0.17 to 0.33] | 0.29 [0.17 to 1.00] | 0.29 [0.08 to 0.50] | 0.25 [0.17 to 0.33] | 0.25 [0.17 to 0.50] | 0.29 [0.08 to 0.50] | 0.33 [0.25 to 0.50]

3. Primary Outcome: Area Under the Curve (AUC0-1.5) of Baseline Adjusted Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*picogram per millilitre (hr*pg/mL)
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
hour*picogram per millilitre (hr*pg/mL) | 4078.68 (2078.89) | 1744.36 (978.81) | 2472.40 (1435.45) | 3635.77 (2069.11) | 1506.23 (541.57) | 2939.31 (1042.03) | 3110.22 (2848.75) | 1999.69 (1329.44)

4. Primary Outcome: Maximum Concentration (Cmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
mg/dL | 138.17 (26.57) | 118.18 (46.46) | 137.50 (42.14) | 130.50 (21.81) | 125.09 (23.81) | 132.82 (30.59) | 123.17 (29.58) | 102.33 (25.63)

5. Primary Outcome: Time to Maximum Concentration (Tmax) of Baseline-Adjusted Glucose
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
hours (hr) | 1.00 [0.67 to 1.50] | 0.67 [0.33 to 1.00] | 1.00 [0.50 to 1.50] | 1.50 [1.00 to 1.50] | 1.00 [0.67 to 1.50] | 1.00 [0.50 to 1.50] | 1.00 [0.67 to 1.50] | 1.00 [0.50 to 1.50]

6. Primary Outcome: Area Under the Effect Concentration Time Curve (AUEC0-1.5) of Baseline-Adjusted Glucose From Time Zero up to 90 Minutes
Time Frame: Pre-dose; 5, 10, 15, 20, 30, 40, 60 and 90 minutes following glucagon administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*mg/dL
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
hr*mg/dL | 145.86 (26.94) | 118.82 (60.73) | 142.38 (51.98) | 132.42 (22.14) | 128.82 (28.45) | 138.12 (35.24) | 126.94 (30.40) | 101.46 (27.38)

7. Secondary Outcome: Nasal and Non-nasal Effects/Symptoms
Description: Symptoms of runny nose, nasal congestion and/or itching, sneezing, watery and/or itchy eyes, redness of eyes, and itching of ears and/or throat were assessed prior to administering glucagon and at 15, 30, 60 and 90 minutes following administration of glucagon. This was done via the "Nasal Non-nasal Score Questionnaire". Each of the 9 symptoms is assigned an integer value from 0 to 3; higher values indicate more severe symptoms (a score of 0 indicates no symptoms). The reported results indicate the cohort median out of a possible maximum value of 27 (summing all 9 questions for each participant and reporting the median/IQR across participants).
Time Frame: Pre-dose;15, 30, 60 and 90 minutes following glucagon administration
Population: All enrolled participants. One participant in the 8 to <12 group withdrew from the study after completion of the 3.0 mg NG visit and did not complete the 2.0 mg NG visit.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 12 | 12 | 6 | 11 | 12 | 12 | 12
units on a scale
  Pre-dose | 0.50 [0.00 to 1.00] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.50] | 0.50 [0.00 to 1.00]
  15 minutes post glucagon administration | 0.00 [0.00 to 1.00] | 1.00 [0.00 to 3.00] | 0.50 [0.00 to 2.00] | 0.00 [0.00 to 1.00] | 3.00 [0.00 to 4.00] | 3.00 [1.00 to 4.50] | 0.00 [0.00 to 0.00] | 2.00 [1.00 to 4.00]
  30 minutes post glucagon administration | 0.00 [0.00 to 1.00] | 1.00 [0.00 to 1.50] | 0.50 [0.00 to 1.50] | 0.00 [0.00 to 1.00] | 2.00 [0.00 to 2.00] | 2.50 [0.50 to 3.50] | 0.00 [0.00 to 0.00] | 1.00 [1.00 to 3.00]
  60 minutes post glucagon administration | 0.00 [0.00 to 0.00] | 0.50 [0.00 to 2.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00] | 0.50 [0.00 to 1.50] | 0.00 [0.00 to 0.00] | 1.00 [0.00 to 2.00]
  90 minutes post glucagon administration | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.50] | 0.00 [0.00 to 0.50] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 0.00] | 1.00 [0.00 to 1.00]

8. Secondary Outcome: Number of Participants Achieving at Least a 25 mg/dL Rise in Blood Glucose Above Nadir Level Within 30 Minutes
Time Frame: Pre-dose; 5, 10, 15, 20, and 30 minutes following glucagon administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
Participants | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12

9. Secondary Outcome: Time to Achieving ≥25 mg/dL Rise in Plasma Glucose Above Nadir Level Within 30 Minutes
Description: Time (in minutes) when all participants experienced a rise in glucose >=25mg/dL. This is an absolute number and is not a calculated statistic. There is no distribution per cohort.
Time Frame: Pre-dose; 5, 10, 15, 20, and 30 minutes following glucagon administration
Population: as for outcome 1
Measure: Number; unit: minutes
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
minutes | 10 | 20 | 15 | 20 | 20 | 15 | 20 | 20

10. Other Pre Specified Outcome: Percentage of Participants With >= 25 mg/dL Rise in Plasma Glucose Within 30 Minutes
Time Frame: Pre-dose; 5, 10,15, 20, and 30 minutes following glucagon administration
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Number analyzed (Participants) | 6 | 11 | 12 | 6 | 11 | 12 | 12 | 12
percentage of participants | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: Through study completion, up to 69 days
Description: Included all participants received at least one dose of glucagon.
Groups:
- 8 to<12 Years Old NG Visit 2.0 mg: NG of 2.0 mg for participants 8 to less than 12 years of age.
Arm/Group | 4 to<8 Years Old IM Glucagon Visit | 4 to<8 Years Old NG Visit 2.0 mg | 4 to<8 Years Old NG Visit 3.0 mg | 8 to <12 Years Old IM Glucagon Visit | 8 to<12 Years Old NG Visit 2.0 mg | 8 to<12 Years Old NG Visit 3.0 mg | 12 to <17 Years Old IM Glucagon Visit | 12 to<17 Years Old NG Visit 3.0 mg
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/12 | 0/12 | 0/6 | 0/11 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/6 | 6/12 | 5/12 | 6/6 | 5/11 | 6/12 | 7/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 to<8 Years Old IM Glucagon Visit (N=6) | 4 to<8 Years Old NG Visit 2.0 mg (N=12) | 4 to<8 Years Old NG Visit 3.0 mg (N=12) | 8 to <12 Years Old IM Glucagon Visit (N=6) | 8 to<12 Years Old NG Visit 2.0 mg (N=11) | 8 to<12 Years Old NG Visit 3.0 mg (N=12) | 12 to <17 Years Old IM Glucagon Visit (N=12) | 12 to<17 Years Old NG Visit 3.0 mg (N=12)
Hypoglycemia (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Experienced a hypoglycemic event after receiving a bolus of insulin with lunch. Received 90 g oral carbohydrates and made a full recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 to<8 Years Old IM Glucagon Visit (N=6) | 4 to<8 Years Old NG Visit 2.0 mg (N=12) | 4 to<8 Years Old NG Visit 3.0 mg (N=12) | 8 to <12 Years Old IM Glucagon Visit (N=6) | 8 to<12 Years Old NG Visit 2.0 mg (N=11) | 8 to<12 Years Old NG Visit 3.0 mg (N=12) | 12 to <17 Years Old IM Glucagon Visit (N=12) | 12 to<17 Years Old NG Visit 3.0 mg (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 2 | 2 | 4 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increase (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 2 | 3 | 1 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 3 | 4 | 5 | 4
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No